CLINICAL TRIAL: NCT05855200
Title: A Phase 3, Open-Label, Randomized Study of Perioperative Dostarlimab Monotherapy Versus Standard of Care in Participants With Untreated T4N0 or Stage III dMMR/MSI-H Resectable Colon Cancer
Brief Title: Study of Perioperative Dostarlimab in Participants With Untreated T4N0 or Stage III dMMR/MSI-H Resectable Colon Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 219606; 2023-503265-27-00 (EU CTIS Number)
Record Dates: First submitted 2023-05-03; First posted 2023-05-11 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Colonic Neoplasms; Neoplasms, Colon
Keywords: JEMPERLI; Dostarlimab; dostarlimab-gxly; TSR-042; GSK4057190A; FOLFOX; CAPEOX; Colon Cancer; Resectable colon cancer; dMMR/MSI; Perioperative; Neoadjuvant; Adjuvant
MeSH Terms: conditions — Colonic Neoplasms | interventions — dostarlimab; Folfox protocol

STUDY DESIGN:
Masking Description: Click here to enter text.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dostarlimab (Experimental): Participants will receive Dostarlimab pre and post surgery
  Interventions: Biological: Dostarlimab
- Standard of Care (SOC) (Active Comparator): Participants will receive SOC (FOLFOX/CAPEOX) or undergo expectant observation post surgery.
  Interventions: Drug: CAPEOX; Drug: FOLFOX

INTERVENTIONS:
Biological: Dostarlimab — Dostarlimab will be administered.
  Arms: Dostarlimab
Drug: CAPEOX — CAPEOX will be administered.
  Arms: Standard of Care (SOC)
Drug: FOLFOX — FOLFOX will be administered.
  Arms: Standard of Care (SOC)

SUMMARY:
The primary purpose of this study is to evaluate the efficacy of perioperative dostarlimab compared with standard of care (SOC) in participants with untreated T4N0 or Stage III (resectable), defective mismatch repair/ microsatellite instability high (dMMR/MSI-H) colon cancer.

ELIGIBILITY:
Inclusion Criteria:

* Has untreated pathologically confirmed colon adenocarcinoma
* Has resectable colon adenocarcinoma defined as clinically T4N0 or Stage III
* Has radiologically evaluable disease
* Has a tumor demonstrating the presence of either dMMR status or MSI-H

Exclusion Criteria:

* Has distant metastatic disease.
* Has received prior medical therapy (chemotherapy, immunotherapy, biologic, or targeted therapy), radiation therapy or surgery for management of the current diagnosis of colon cancer
* Has a tumor that, in the investigator's judgment is causing symptomatic bowel obstruction or otherwise requires urgent/emergent surgery at the time of screening. Participants with a history of colonic obstruction are eligible after obstruction is relieved by a diverting stoma (defunctioning ileostomy or colostomy). Patients with a history of colonic obstruction in the context of current colon cancer diagnosis and treated with colonic stents are not eligible.
* Has undergone any major surgical procedure, open biopsy, or experienced significant traumatic injury within 28 days prior to randomization
* Has any history of interstitial lung disease or pneumonitis and/or history of radiation induced enteritis.
* Has cirrhosis or current unstable liver or biliary disease per investigator assessment defined by the presence of ascites, encephalopathy, coagulopathy, hypoalbuminemia, esophageal/gastric varices, or persistent jaundice
* Has a history of allogenic stem cell transplantation or organ transplantation
* Is receiving any other anticancer or experimental therapy. No other experimental therapies (including but not limited to chemotherapy, radiation, hormonal treatment, antibody therapy, immunotherapy, gene therapy, vaccine therapy, or other experimental drugs) of any kind are permitted while the participant is receiving study intervention
* Is pregnant, breastfeeding, or expecting to conceive children within the projected duration of the study
* Has a history of severe allergic and/or anaphylactic reactions to chimeric, human or humanized antibodies, fusion proteins, or known allergies to dostarlimab, or its excipients, or any components of FOLFOX or CAPEOX

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 892 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2029-03-19 (Estimated); Study Completion 2031-03-27 (Estimated)

PRIMARY OUTCOMES:
Event-free Survival (EFS) Assessed by Blinded Independent Central Review (BICR) | Up to approximately 5 years
  EFS is defined as the time from randomization to either disease recurrence or death due to any cause or treatment related toxicity that results in the participant not being suitable for surgery

SECONDARY OUTCOMES:
Overall Survival (OS) | Up to approximately 5 years
  OS is defined as time from randomization to death from any cause
Number of Participants with Pathological Response | Up to approximately 5 years
  Pathological response will be categorized as a complete pathologic response, major pathologic response, partial pathologic response, or negligible pathologic response.
Event-free Survival (EFS) assessed by local assessment | Up to approximately 5 years
  EFS is defined as the time from randomization to either disease recurrence or death due to any cause or treatment related toxicity that results in the participant not being suitable for surgery
Number of Participants with treatment emergent adverse events (AEs), serious adverse events (SAEs), Immune-mediated Adverse Event (imAEs), AEs leading to death and AEs leading to discontinuation of study treatment | Up to approximately 5 years
Number of Participants with AEs and SAEs by Severity | Up to approximately 5 years
Serum Concentration of Dostarlimab | Predose and End of Infusion (EoI) of Cycle 1 and EoI of Cycle 2 to Cycle 10 (each cycle is of 21 days)
Serum Concentration of Dostarlimab at End of Infusion (C-EoI) | End of Infusion (EoI) of Cycle 1 to Cycle 10 (each cycle is of 21 days)
Serum Predose trough concentration (Ctrough) of Dostarlimab | Predose of Cycle 1 to Cycle 10 (each cycle is of 21 days)
Number of Participants with Anti-Drug Antibodies against Dostarlimab | Up to approximately 5 years

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (209):
- United States (34):
  - GSK Investigational Site, Tucson, Arizona
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, New Haven, Connecticut
  - GSK Investigational Site, Washington D.C., District of Columbia
  - GSK Investigational Site, Deerfield Beach, Florida
  - GSK Investigational Site, Fort Lauderdale, Florida
  - GSK Investigational Site, Marietta, Georgia
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Naperville, Illinois
  - GSK Investigational Site, Westwood, Kansas
  - GSK Investigational Site, Lexington, Kentucky
  - GSK Investigational Site, Louisville, Kentucky
  - GSK Investigational Site, Baton Rouge, Louisiana
  - GSK Investigational Site, Bethesda, Maryland
  - GSK Investigational Site, Ann Arbor, Michigan
  - GSK Investigational Site, Detroit, Michigan
  - GSK Investigational Site, Minneapolis, Minnesota
  - GSK Investigational Site, Joplin, Missouri
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Grand Island, Nebraska
  - GSK Investigational Site, Omaha, Nebraska
  - GSK Investigational Site, Lebanon, New Hampshire
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, The Bronx, New York
  - GSK Investigational Site, Durham, North Carolina
  - GSK Investigational Site, Akron, Ohio
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Sioux Falls, South Dakota
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Richmond, Virginia
  - GSK Investigational Site, Appleton, Wisconsin
- Argentina (8):
  - GSK Investigational Site, Buenos Aires
  - GSK Investigational Site, Capital Federal
  - GSK Investigational Site, Ciudad Autonoma de Buenos Aire
  - GSK Investigational Site, Córdoba
  - GSK Investigational Site, Mar del Plata
  - GSK Investigational Site, Rosario
  - GSK Investigational Site, San Miguel de Tucumán
  - GSK Investigational Site, Santa Fe
- Australia (5):
  - GSK Investigational Site, Newcastle, New South Wales
  - GSK Investigational Site, St Leonards, New South Wales
  - GSK Investigational Site, Woolangabba, Queensland
  - GSK Investigational Site, Heidelberg, Victoria
  - GSK Investigational Site, Melbourne, Victoria
- Belgium (7):
  - GSK Investigational Site, Aalst
  - GSK Investigational Site, Brussels
  - GSK Investigational Site, Edegem
  - GSK Investigational Site, Ghent
  - GSK Investigational Site, Leuven
  - GSK Investigational Site, Liège
  - GSK Investigational Site, Roeselare
- Brazil (11):
  - GSK Investigational Site, Barretos
  - GSK Investigational Site, Belém
  - GSK Investigational Site, Campo Grande
  - GSK Investigational Site, Lages
  - GSK Investigational Site, Natal
  - GSK Investigational Site, Porto Alegre
  - GSK Investigational Site, Salvador
  - GSK Investigational Site, São José do Rio Preto
  - GSK Investigational Site, São Paulo
  - GSK Investigational Site, Teresina
  - GSK Investigational Site, Vitória
- Canada (5):
  - GSK Investigational Site, Edmonton, Alberta
  - GSK Investigational Site, Halifax, Nova Scotia
  - GSK Investigational Site, Ottawa, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Montreal, Quebec
- China (20):
  - GSK Investigational Site, Beijing
  - GSK Investigational Site, Changchun
  - GSK Investigational Site, Changsha
  - GSK Investigational Site, Chengdu
  - GSK Investigational Site, Chongqing
  - GSK Investigational Site, Guangzhou
  - GSK Investigational Site, Hangzhou
  - GSK Investigational Site, Harbin
  - GSK Investigational Site, Jinan
  - GSK Investigational Site, Kunming
  - GSK Investigational Site, Meizhou
  - GSK Investigational Site, Nanchang
  - GSK Investigational Site, Shanghai
  - GSK Investigational Site, Shenzhen
  - GSK Investigational Site, Taiyuan
  - GSK Investigational Site, Tianjin
  - GSK Investigational Site, Wuhan
  - GSK Investigational Site, Xiamen
  - GSK Investigational Site, Yangzhou
  - GSK Investigational Site, Zhengzhou
- Czechia (3):
  - GSK Investigational Site, Hradec Králové
  - GSK Investigational Site, Nový Jičín
  - GSK Investigational Site, Prague
- Estonia (2):
  - GSK Investigational Site, Tallinn
  - GSK Investigational Site, Tartu
- Finland (3):
  - GSK Investigational Site, Helsinki
  - GSK Investigational Site, Tampere
  - GSK Investigational Site, Turku
- France (11):
  - GSK Investigational Site, Lyon
  - GSK Investigational Site, Marseille
  - GSK Investigational Site, Nantes
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Pessac
  - GSK Investigational Site, Rennes
  - GSK Investigational Site, Rouen
  - GSK Investigational Site, Saint-Priest-en-Jarez
  - GSK Investigational Site, Suresnes
  - GSK Investigational Site, Toulouse
  - GSK Investigational Site, Villejuif
- Germany (7):
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Düsseldorf
  - GSK Investigational Site, Frankfurt
  - GSK Investigational Site, Halle
  - GSK Investigational Site, Lübeck
  - GSK Investigational Site, Mannheim
  - GSK Investigational Site, München
- Greece (2):
  - GSK Investigational Site, Athens
  - GSK Investigational Site, Thessaloniki
- India (6):
  - GSK Investigational Site, Bengaluru, Karnataka
  - GSK Investigational Site, Ludhiana, Punjab
  - GSK Investigational Site, Belagavi
  - GSK Investigational Site, Hyderabad
  - GSK Investigational Site, Nashik
  - GSK Investigational Site, Pune
- Italy (9):
  - GSK Investigational Site, Cagliari
  - GSK Investigational Site, Genova
  - GSK Investigational Site, Milan
  - GSK Investigational Site, Napoli
  - GSK Investigational Site, Padua
  - GSK Investigational Site, Pisa
  - GSK Investigational Site, Reggio Emilia
  - GSK Investigational Site, Roma
  - GSK Investigational Site, Rozzano MI
- Japan (12):
  - GSK Investigational Site, Aichi
  - GSK Investigational Site, Chiba
  - GSK Investigational Site, Fukuoka
  - GSK Investigational Site, Hokkaido
  - GSK Investigational Site, Hyōgo
  - GSK Investigational Site, Ibaraki
  - GSK Investigational Site, Kanagawa
  - GSK Investigational Site, Kyoto
  - GSK Investigational Site, Okayama
  - GSK Investigational Site, Osaka
  - GSK Investigational Site, Shizuoka
  - GSK Investigational Site, Tokyo
- Mexico (6):
  - GSK Investigational Site, DF
  - GSK Investigational Site, Guadalajara
  - GSK Investigational Site, Mexico City
  - GSK Investigational Site, Oaxaca City
  - GSK Investigational Site, San Pedro Garza García
  - GSK Investigational Site, Tijuana
- Netherlands (4):
  - GSK Investigational Site, Breda
  - GSK Investigational Site, Maastricht
  - GSK Investigational Site, Nijmegen
  - GSK Investigational Site, Utrecht
- Norway (6):
  - GSK Investigational Site, Bergen
  - GSK Investigational Site, Kristiansand
  - GSK Investigational Site, Lrenskog
  - GSK Investigational Site, Oslo
  - GSK Investigational Site, Stavanger
  - GSK Investigational Site, Tromsø
- GSK Investigational Site, Punta Pacifica Panama City Panama, Panama
- Poland (2):
  - GSK Investigational Site, Bydgoszcz
  - GSK Investigational Site, Warsaw
- Portugal (3):
  - GSK Investigational Site, Almada
  - GSK Investigational Site, Coimbra
  - GSK Investigational Site, Lisbon
- South Korea (3):
  - GSK Investigational Site, Daegu
  - GSK Investigational Site, Gyeonggi-do
  - GSK Investigational Site, Seoul
- Spain (18):
  - GSK Investigational Site, Badajoz
  - GSK Investigational Site, BaracaldoVizcaya
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Córdoba
  - GSK Investigational Site, Donostia / San Sebastian
  - GSK Investigational Site, Elche Alicante
  - GSK Investigational Site, Granada
  - GSK Investigational Site, Jaén
  - GSK Investigational Site, L'Hospitalet de Llobrega
  - GSK Investigational Site, Las Palmas de Gran Canar
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Málaga
  - GSK Investigational Site, Oviedo
  - GSK Investigational Site, Pamplona
  - GSK Investigational Site, Santander
  - GSK Investigational Site, Seville
  - GSK Investigational Site, Valencia
  - GSK Investigational Site, Zaragoza
- Sweden (6):
  - GSK Investigational Site, Eskilstuna
  - GSK Investigational Site, Gothenburg
  - GSK Investigational Site, Linköping
  - GSK Investigational Site, Malmo
  - GSK Investigational Site, Stockholm
  - GSK Investigational Site, Uppsala
- Taiwan (4):
  - GSK Investigational Site, Kaohsiung City
  - GSK Investigational Site, Tainan
  - GSK Investigational Site, Taipei
  - GSK Investigational Site, Taoyuan District
- Turkey (Türkiye) (2):
  - GSK Investigational Site, Ankara
  - GSK Investigational Site, Istanbul
- United Kingdom (9):
  - GSK Investigational Site, Birmingham
  - GSK Investigational Site, Chelmsford
  - GSK Investigational Site, Cheltenham
  - GSK Investigational Site, Edinburgh
  - GSK Investigational Site, Hull
  - GSK Investigational Site, Leeds West Yorkshire
  - GSK Investigational Site, London
  - GSK Investigational Site, Manchester
  - GSK Investigational Site, Sutton

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to anonymized individual patient-level data (IPD) and related study documents of the eligible studies via the Data Sharing Portal. Details on GSK's data sharing criteria can be found at: https://www.gsk.com/en-gb/innovation/trials/data-transparency/
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk.com/en-gb/innovation/trials/data-transparency/

REFERENCES:
- [Derived] Starling N, Elez E, Strickler JH, Benson A, Oki E, Mendez G, Ferreiro R, Lau YL, Kawazoe A, Tian M, Campbell N, Cohen DN, Edwards K, Stjepanovic N, Seligmann JF. A Phase III study of perioperative dostarlimab in patients with dMMR/MSI-H resectable colon cancer: AZUR-2 study design. Future Oncol. 2026 Jan;22(2):137-145. doi: 10.1080/14796694.2025.2606910. Epub 2026 Jan 6. PMID 41492912